CLINICAL TRIAL: NCT05203679
Title: A Phase 1/2/3 Open-label Study to Evaluate the Safety, Tolerability and Efficacy of an Adeno-associated Virus Vector Containing an Expression Cassette of the Human Factor IX Transgene (BBM-H901) Injection in Patients With Hemophilia B
Brief Title: Evaluation of the Safety and Efficacy of Hemophilia B Gene Therapy Drug
Status: Active, not recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Shanghai Xinzhi BioMed Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BBM001-CLN1001
Record Dates: First submitted 2021-12-29; First posted 2022-01-24 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: Hemophilia B
Keywords: Hemophilia B;gene therapy;Adeno-Associated Virus
MeSH Terms: conditions — Hemophilia B

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Arm of BBM-H901 (Experimental): Single-dose treatment
  Interventions: Genetic: Single dose intravenous injection of BBM-H901

INTERVENTIONS:
Genetic: Single dose intravenous injection of BBM-H901 — Single dose intravenous infusion of BBM-H901, an adeno-associated virus (AAV) vector derived from recombinant DNA techniques to contain an expression cassette of the human factor IX (hFIX) transgene in liver.

SUMMARY:
This is a multi-center, Phase 1/2/3, single-arm, open-label, single-dose treatment clinical study to evaluate the safety, tolerability and efficacy of BBM-H901 injection in Hemophilia B subjects with ≤2 International unit per deciliter (IU/dl) residual factor IX (FIX) levels.

BBM-H901 is an adeno-associated virus (AAV) vector derived from recombinant DNA techniques to contain an expression cassette of the human factor IX (hFIX) transgene and raises circulating levels of endogenous FIX.

ELIGIBILITY:
Inclusion Criteria of Phase 1/2/3:

1. Males ≥ 18 years of age;
2. Have hemophilia B with ≤2 IU/dL (≤2 %) endogenous FIX activity levels;
3. Have had ≥100 prior exposure days (EDs) to any recombinant and/or plasma-derived FIX protein products based on historical data from the subjects' records/histories;
4. Have had bleeding events and/or injected with FIX protein products (including recombination and plasma source) during the last 12 weeks documented in the subjects' medical records;
5. Have no prior history of hypersensitivity or anaphylaxis associated with any FIX or IV immunoglobulin administration;
6. Agree to use a reliable barrier contraception method from the beginning of signing the informed consent to 52 weeks after administration.

Exclusion Criteria of Phase 1/2/3:

1. Being positive for hepatitis B surface antigen (HBsAg) or hepatitis B virus-DNA (HBV-DNA). Being positive for hepatitis C virus antibody (HCV-Ab) or hepatitis C virus RNA (HCV-RNA). Subjects with medical history of hepatitis B or C can be regarded as negative only when 2 required samplings are conducted at least 3 months apart and both test results of indicators aforementioned are negative, i.e. subjects with natural clearance and anti-viral therapy clearance for hepatitis B or C are eligible;
2. Have potential liver diseases, such as previous diagnosis of portal hypertension, splenomegaly, hepatic encephalopathy or liver fibrosis (fibrosis stage ≥ 3); nodules or cysts were found by B ultrasound, or elevated alpha-fetoprotein was detected by laboratory tests. Subjects who are not eligible for the study if the abnormalities are clinically significant regarding to the medical judgement of the investigator;
3. HIV positive patients;
4. Have participated in a previous gene therapy research trial before screening, or in a clinical study with an investigational drug within 5 half-life of the investigational product, whichever is longer;
5. Have alcohol or drug dependence, or cannot stop drinking throughout the study;
6. Any concurrent clinically significant major disease or condition that the investigator deems unsuitable for participation in the study.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2021-12-30 (Actual); Primary Completion 2024-04-16 (Actual); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Phase 1/2: The incidence of dose limiting toxicity (DLT) events | 10 weeks post-infusion
  To access the numbers of DLT events determined by the Safety Data Review Committee (SRC) in DLT observation period after BBM-H901 injection infusion.
Phase 1/2: The incidence of adverse events (AEs) and serious adverse events (SAEs) | 10 weeks post-infusion
  To assess the safety of BBM-H901 Injection by AEs and SAEs.
Phase 1/2: Changes in liver function | 10 weeks post-infusion
  To assess changes in liver function before and after treatment, including alanine aminotransferase (ALT) and aspartate aminotransferase (AST).
Phase 3: Annualized bleeding rate (ABR) | 52 weeks post-infusion
  To assess ABR, including spontaneous bleeding and traumatic bleeding after administration.

SECONDARY OUTCOMES:
Phase 1/2: Changes in liver function | 52 weeks post-infusion
  To assess changes in liver function before and after treatment, including alanine aminotransferase (ALT) and aspartate aminotransferase (AST).
Phase 1/2/3: Mean FIX Padua Activity Level | 52 weeks post-infusion
  Measurement of mean FIX Padua activity levels over the 52-week period following BBM-H901 injection.
Phase 1/2/3: Other FIX Protein Product Usage | 52 weeks post-infusion
  Number and total volume of infusions of exogenous FIX protein products (recombinant or plasma-derived) administered within 52 weeks post-BBM-H901 injection.
Phase 1/2/3: Target Joint Count | 52 weeks post-infusion
  Number of target joints recorded within 52 weeks post-BBM-H901 injection.
Phase 1/2/3: Joint Bleeding Episodes | 52 weeks post-infusion
  Total number of joint bleeding events occurring within 52 weeks post-BBM-H901 injection.
Phase 1/2/3: Bleeding-Free Subjects | 52 weeks post-infusion
  Proportion of subjects experiencing no bleeding events within 52 weeks post-BBM-H901 injection.
Phase 1/2/3: Adverse Event Incidence | 52 weeks post-infusion
  Incidence of adverse events (AEs) and serious adverse events (SAEs) within 52 weeks post-BBM-H901 injection.
Phase 1/2/3: FIX Inhibitor Incidence | 52 weeks post-infusion
  Incidence of FIX inhibitors measured by Bethesda or Nijmegen-Bethesda assays within 52 weeks post-BBM-H901 injection.
Phase 1/2/3: AAV Vector Shedding | 52 weeks post-infusion
  Changes in AAV vector shedding in plasma, urine, semen, saliva, and PBMCs within 52 weeks post-BBM-H901 injection.

CONTACTS AND LOCATIONS:
Overall Officials: Lei Zhang, MD, Study Chair — Institute of Hematology & Blood Diseases Hospital Chinese Academy of Medical Sciences & Peking Union Medical College; Caifeng Yang, Master, Study Director — Shanghai Xinzhi BioMed Co., Ltd.
Locations (9):
- China (9):
  - Anhui Provincial Hospital, Hefei, Anhui
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - Nanfang Hospital Southern Medical University, Guangzhou, Guangdong
  - The Second People's Hospital of Shenzhen, Shenzhen, Guangdong
  - North China University of Science and Technology Affiliated Hospital, Tangshan, Hebei
  - Henan Cancer Hospital, Zhengzhou, Henan
  - The Second Hospital of Shanxi Medical University, Taiyuan, Shanxi
  - Institute of Hematology & Blood Diseases Hospital Chinese Academy of Medical Sciences & Peking Union Medical College, Tianjin, Tianjin Municipality
  - The second Affiliated Hospital of Kunming Medical University, Kunming, Yunnan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Xue F, Ju M, Zhu T, Zhou Z, Sun J, Yang L, Yan Z, Zhou H, Du X, Zheng C, Zheng J, Wu X, Du Z, Jiang W, Yang C, Xiao X, Liu W, Yang R, Zhang L. Factor IX-Padua AAV gene therapy in hemophilia B: phases 1/2 and 3 trials. Nat Med. 2026 Jan;32(1):93-102. doi: 10.1038/s41591-025-04012-y. Epub 2025 Nov 20. PMID 41266685